CLINICAL TRIAL: NCT03049215
Title: Lumen Apposing Metal Stents vs Lumen Apposing Metal Stent Plus Double Pigtail Stent for Endoscopic Drainage of Pancreatic Fluid Collections: a Randomized Controlled Trial
Brief Title: Lumen Apposing Metal Stents vs Lumen Apposing Metal Stent Plus Double Pigtail Stent for Endoscopic Drainage
Acronym: Axios
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to low/difficulty enrollment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Yachimski, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170247
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Pseudocyst
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either: LAMS alone and undergo EUS-guided transmural placement of an Axios stent with a 15 mm luminal diameter or LAMS plus double pigtail stent and undergo EUS-guided transmural placement of a single Axios stent with a 15 mm luminal diameter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Lumen Apposing Metal Stent (LAMS) (Active Comparator): Subjects randomized to LAMS alone will undergo EUS-guided transmural placement of an Axios stent with a 15 mm luminal diameter.
  Interventions: Device: Lumen Apposing Metal Stent (LAMS)
- LAMS plus double pigtail stent (Active Comparator): Subjects randomized to LAMS plus double pigtail stent will undergo EUS-guided transmural placement of a single Axios stent with a 15 mm luminal diameter. Following this, wire access across the stent lumen will be achieved using a 0.035 inch hydrophilic guidewire, and a double pigtail plastic biliary stent (6 French, 7 French, or 10 French at the discretion of the endoscopist) will be deployed over the wire.
  Interventions: Device: LAMS plus double pigtail stent

INTERVENTIONS:
Device: Lumen Apposing Metal Stent (LAMS) — The AXIOS Stent and Electrocautery-Enhanced Delivery System is an endoscopic device designed to enable the ultrasound trained interventional endoscopist to deliver a transenteric stent between the gastrointestinal tract and a pancreatic pseudocyst.
  Other Names: Axios Stent
  Arms: Lumen Apposing Metal Stent (LAMS)
Device: LAMS plus double pigtail stent — The AXIOS Stent and Electrocautery-Enhanced Delivery System is an endoscopic device designed to enable the ultrasound trained interventional endoscopist to deliver a transenteric stent between the gastrointestinal tract and a pancreatic pseudocyst. The double pigtail stent is a routinely used plastic biliary stent.
  Arms: LAMS plus double pigtail stent

SUMMARY:
The study hypothesis is that placement of LAMS plus an overlapping double pigtail stent for endoscopic transmural drainage of PFCs with solid debris will result in improved drainage and require fewer endoscopic interventions compared to placement of LAMS alone.

DETAILED DESCRIPTION:
The study hypothesis is that placement of LAMS plus an overlapping double pigtail stent for endoscopic transmural drainage of PFCs with solid debris will result in improved drainage and require fewer endoscopic interventions compared to placement of LAMS alone.

Adult patients with symptomatic pancreatic fluid collections who are scheduled to undergo EUS-guided drainage of PFCs with LAMS placement will be eligible for study participation. The initial portion of this procedure consists of diagnostic EUS for imaging and assessment of the PFC. This EUS examination is able to distinguish the relative liquid and solid components of PFCs, detail which may not be evident by CT imaging. Adult patients with PFCs consisting of >30% solid component as assessed at the time of EUS will be eligible for randomization. This threshold was selected as the enrollment criteria in order to select patients with a significant solid necrotic component to the lesion, as prior study of patients undergoing LAMS placement for drainage of PFCs have used >70% fluid content as the definition for a PFC with predominantly liquid contents.

Allocation to study arm will be determined by the contents of sealed envelope. Subjects randomized to LAMS alone will undergo EUS-guided transmural placement of an Axios stent with a 15 mm luminal diameter. The choice of transgastric or transduodenal LAMS placement will be at the discretion of the endoscopist and contingent upon PFC location and window relative to the EUS transducer. Subjects randomized to LAMS plus double pigtail stent will undergo EUS-guided transmural placement of a single Axios stent with a 15 mm luminal diameter; following this, wire access across the stent lumen will be achieved using a 0.035 inch hydrophilic guidewire, and a double pigtail plastic biliary stent (6 French, 7 French, or 10 French at the discretion of the endoscopist) will be deployed over the wire. The use of fluoroscopy for stent deployment will be at the discretion of the endoscopist.

The primary end point: Greater than 50% decrease in size of PFC (in mm), compared to pre-intervention size (in mm), on cross-sectional computed tomography (CT) imaging at 30 days following stent placement. This was selected as the primary outcome in order to maintain consistency with the primary outcomes of a prior multicenter study of LAMS placement for PFCs.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients between the ages of 18 and 80
* Must be presenting with symptomatic pancreatic fluid collections
* Scheduled to undergo endoscopic ultrasound (EUS)-guided drainage of PFCs with LAMS placement at Vanderbilt Medical Center as part of routine care
* Willing and able to give informed consent

Exclusion Criteria:

* Unwilling/unable to give informed consent
* Patients with PFCs consisting of < 30% solid component as assessed at the time of EUS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yachimski, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from patient population at the Vanderbilt Digestive Disease Center. One participant was enrolled on November 6, 2017, however they were not randomized. A second participant was enrolled in June 2018. No other participants were enrolled.
Pre-assignment Details: 2 participants were enrolled (signed consent). However, only 1 participant was randomized and completed the study.
Period: Overall Study
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was ever enrolled on the study, and this participant was randomized to the Lumen Apposing Metal Stent (LAMS) arm. No participants were randomized to the LAMS plus double pigtail stent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (0) |  | 62 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Pancreatic Fluid Collection (PFC)
Description: Greater than 50% decrease in size of PFC (in mm) compared to pre-intervention size (in mm) as measured on cross-sectional computed tomography (CT) imaging
Time Frame: 30 days following placement of stent
Population: No participants were randomized to the LAMS plus double pigtail stent arm
Measure: Number; unit: percentage of decrease
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent
Number analyzed (Participants) | 1 | 0
percentage of decrease | 64 |

2. Secondary Outcome: Clinical Success Rate for Draining of Pancreatic Fluid Collection (PFC)
Description: Clinical success for drainage of PFC, defined as complete resolution of PFC on follow-up computed tomography (CT) imaging and stent removal within 3 months
Time Frame: 3 months
Population: No participants were randomized to LAMS plus double pigtail stent
Measure: Count of Participants; unit: Participants
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

3. Secondary Outcome: Number of Endoscopic Interventions Required for Resolution of PFC Prior to Stent Removal
Description: Number of endoscopic interventions required for resolution of Pancreatic Fluid Collection (PFC) prior to stent removal
Time Frame: 3 months
Population: No participants were randomized to the LAMS plus double pigtail stent arm
Measure: Number; unit: number of interventions
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent
Number analyzed (Participants) | 1 | 0
number of interventions | 2 |

4. Secondary Outcome: Incidence of Hospital Readmissions Following Initial Endoscopic Intervention and Prior to Resolution of Pancreatic Fluid Collection Stent Removal
Description: Incidence of hospital readmissions following initial endoscopic intervention and prior to resolution of Pancreatic Fluid Collection (PFC) stent removal
Time Frame: 3 months
Population: No participants were randomized to the LAMS plus double pigtail stent arm
Measure: Number; unit: event
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent
Number analyzed (Participants) | 1 | 0
event | 1 |

5. Secondary Outcome: Incidence of Surgical or Percutaneous Radiologic Intervention for PFC Following Initial Endoscopy Intervention
Description: Incidence of surgical or percutaneous radiologic intervention for Pancreatic Fluid Collection (PFC) following initial endoscopy intervention
Time Frame: 3 months
Population: No participants were randomized to the LAMS plus double pigtail stent arm
Measure: Number; unit: event
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent
Number analyzed (Participants) | 1 | 0
event | 0 |

6. Secondary Outcome: Incidence of Early (<30 Days) Endoscopic Reintervention
Description: Incidence of early (<30 days) endoscopic reintervention following initial endoscopic intervention
Time Frame: 30 days
Population: No participants were randomized to the LAMS plus double pigtail stent arm
Measure: Number; unit: event
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent
Number analyzed (Participants) | 1 | 0
event | 1 |

ADVERSE EVENTS:
Time Frame: 18 months
Description: Definition of adverse event and/or serious adverse event did not differ from the clinicaltrials.gov definitions.
Arm/Group | Lumen Apposing Metal Stent (LAMS) | LAMS Plus Double Pigtail Stent
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Terminated due to low/difficulty enrollment. Only one participant was randomized. As a result, originally planned analysis was not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT03049215/Prot_SAP_001.pdf